CLINICAL TRIAL: NCT02443948
Title: Circulating Cell-free Tumor DNA in the Plasma of Patients With Gastrointestinal Stromal Tumors (GIST): Detection and Correlation With Disease Status Assessed by Conventional Technique. Prospective Observational Study
Brief Title: Circulating Cell-free Tumor DNA in the Plasma of Patients With Gastrointestinal Stromal Tumors (GIST)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: cf-DNA GIST
Record Dates: First submitted 2015-03-19; First posted 2015-05-14 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cf-DNA blood samples will be collected in EDTA tubes during the routine blood test.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- adjuvant/follow up setting
  Interventions: Other: Vena puncture for blood collection
- neo-adjuvant setting
  Interventions: Other: Vena puncture for blood collection
- advanced disease
  Interventions: Other: Vena puncture for blood collection

INTERVENTIONS:
Other: Vena puncture for blood collection — Cf-DNA blood samples will be collected in EDTA tubes (20 ml) during the routine blood test

SUMMARY:
This observational study is proposed to evaluate if the trend in the levels of cf-DNA evaluated on a sample of peripheral blood may be related to different clinical behaviors of the disease monitored by radiological investigations conducted.

DETAILED DESCRIPTION:
Demetri and colleagues presented, at the AACR and ASCO Annual Meeting 2013, an exploratory analysis to assess GIST genotypes on patients in the GRID study. Mutations in the KIT gene were detected in 58 percent of the blood samples compared with 66 percent of the tumor tissue samples (31). However, when focusing their analysis on secondary KIT mutations, which are the mutations that drive resistance to targeted therapies like imatinib and sunitinib, the researchers found mutations in 47 percent of blood samples compared with only 12 percent of tissue samples. In addition, nearly half of blood samples in which secondary KIT mutations were found, harbored multiple secondary mutations. Therefore, cf-DNA may become an efficient marker of mutational GIST status and disease itself.

On this basis, this trial aims to evaluate whether tumor DNA carrying mutations (for KIT, PDGFRα, BRAF, RAS, SDH) can be detected and quantified in the plasma of patients with GISTs, either with active disease or during follow-up, and whether detection can be correlated with the disease status.

ELIGIBILITY:
* Male or female patients aged >= 18 years
* Histologically confirmed diagnosis of GIST of any anatomical location either by biopsy or surgical specimen
* Available archival tumor tissue
* Signed informed consent form

Exclusion Criteria:

* Impossibility to ensure adequate clinical and serum sample follow-up
* Serious psychiatric disease that precludes informed consent or limits compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes adult patients with histologically confirmed GIST, either with active disease or in follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of change in cf-DNA levels with disease status in GIST patients harboring specific DNA mutations | baseline, every 12 weeks, up to 2 years
  To assess the correlation of change in cf-DNA levels with disease status evaluated according to RECIST criteria v 1.1

SECONDARY OUTCOMES:
Clearance of cf-DNA levels after surgery in GIST patients harboring specific DNA mutations | the day before surgery, every 12 weeks, up to 2 years
  To evaluate the time (half-life esteem) of cf-DNA levels clearance after definitive surgery
Detection of secondary mutations in KIT, PDGFRα and/or other genes | baseline, every 12 weeks, up to 2 years
  To evaluate the possibility to detect secondary mutations in KIT, PDGFRα and/or other genes
Correlation of cf-DNA levels with overall survival (OS) | baseline and up to 2 years
  To evaluate the correlation between cf-DNA levels and overall survival (time from the date of enrollment to date of death or to the date being censored at two years, whichever occurs first)
Correlation of detection of secondary mutations in KIT, PDGFRα and/or other genes with radiological disease progression | baseline, every 12 weeks, up to 2 years
  To correlate the detection of secondary mutations in KIT, PDGFRα and/or other genes with radiological disease progression according to RECIST criteria v 1.1
Correlation of the level of cf-DNA related to disease status in GIST patients harboring specific DNA mutations | baseline, every 12 weeks, up to 2 years
  To assess if the cf-DNA levels are related to disease status detected according to Choi criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione del Piemonte per l'Oncologia, Candiolo, TO, Italy